CLINICAL TRIAL: NCT05543655
Title: Impact of Simulation-Based Training on the Safety of Medication Administration
Acronym: SIM-SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC22_0241
Record Dates: First submitted 2022-09-05; First posted 2022-09-16 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Health Knowledge, Attitudes, Practice; Nurse Training; Simulation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: 10 training courses including 4 nurses each are scheduled, i.e. 40 inclusions. The nurses will benefit from two half-days of simulation training three-months apart, dealing with the safety of medication administration. The training will include a high-fidelity scenario whose events will be adapted to medication administration in conventional care services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- simulated (Experimental): The 'Simulation training', using high fidelity simulation with a simulated patient, is composed of 2 training sessions of 3 hours each. The training will include a high-fidelity scenario whose events will be adapted to medication administration in conventional care services. This scenario is developed by a multidisciplinary team of healthcare professionals, experts in simulation and risk management
  Interventions: Other: high fidelity simulation

INTERVENTIONS:
Other: high fidelity simulation — Each half-day training session will begin with a reminder of the context and general objectives of the training. Nurses will complete the self-assessment and knowledge tests.
  The nurses, each in turn, will start the scenario and will immediately assess the workload felt, by the Nasa-TLX grid. During these high-fidelity simulation sessions, an "error cart" workshop will allow all the other nurses to summon up their knowledge on safety tools upstream of the administration procedure.
  The session begins with a briefing and ends with a debriefing.

SUMMARY:
Task interruption is part of professional life. The healthcare world is not exempt from this phenomenon. Task interruptions lead to errors and increase the risks in managing patients.

Medication administration is the critical step, in that it is the final step to stop medication errors produced upstream. It therefore requires the full attention of any healthcare professional.

In the field of health, simulation has become an innovative educational tool allowing experiential learning and reflective practice.

The general aim of this study is to objectivize the value of simulation-based training as regards medication administration when task interruptions occur.

ELIGIBILITY:
Inclusion Criteria:

* Nurses from conventional medical and surgical departments participating in the training
* people agreeing to participate in the study

Exclusion Criteria:

* Person refusing the processing of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
The effectiveness of simulation-based training on safe drug administration for nurses in conventional services in terms of the number of good steps achieved among the 10 proposed by the HAS | three month
  Difference between the two assessments of the number of good steps performed during the process

CONTACTS AND LOCATIONS:
Locations (1):
- Simulation center All'Sims; University Hospital of Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No